CLINICAL TRIAL: NCT01556958
Title: Prospective Comparative Study of WheezeRATE™ (Wz%) Readings With Spirometry, Symptoms, and Auscultatory Findings in Children With Wheezing.
Brief Title: WheezoMeter® Correlation Study
Status: Terminated | Type: Observational
Why Stopped: Device revised
Sponsor: iSonea (Industry)
Responsible Party: Sponsor
Other Study IDs: iS-2012-Wz
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Asthma; Bronchiolitis
MeSH Terms: conditions — Asthma; Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Active Wheezing - age 5-12
- Active Wheezing - under age 5
- No Wheezing

SUMMARY:
The primary goal of the study is to more firmly establish correlations between WheezeRate(Wz%) and other parameters used to assess wheezing and asthma including spirometry, provider's auscultation, and symptoms at the time of Wz% measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients <= 12 years of age who have wheezing at the time of study as confirmed by the physicians' auscultation.

Control:

* Patients <= 12 years of age without history of asthma or other pulmonary conditions, and who are without wheezing on physical exam.

Exclusion Criteria:

* Medical problems that would contraindicate Wz% measurement.

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric Specialty Clinic
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 1, Folsom, California, United States